CLINICAL TRIAL: NCT06578507
Title: Pharmacokinetics, Efficacy and Safety of Twice Daily Dosing Regimen of Hydroxycarbamide Dispersible Tablets in Children With Sickle Cell Disease: a Single-group, Non-randomised, Open-label Study (KID-BID)
Brief Title: Pharmacokinetics, Efficacy and Safety of Twice Daily Dosing Regimen of Hydroxycarbamide Dispersible Tablets in Children With Sickle Cell Disease
Acronym: KID-BID
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Theravia (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SIK-FR-24-1
Record Dates: First submitted 2024-08-22; First posted 2024-08-29 (Actual); Last update posted 2025-09-17 (Actual); Status verified 2025-09

CONDITIONS: Sickle Cell Disease
Keywords: Hydroxycarbamide; Pharmacokinetic
MeSH Terms: conditions — Anemia, Sickle Cell | interventions — Hydroxyurea

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Hydroxycarbamide Pediatric dispersible tablet (Experimental): Hydroxycarbamide Pediatric dispersible tablet will be administered twice daily during 12 months.
  Interventions: Drug: Hydroxycarbamid

INTERVENTIONS:
Drug: Hydroxycarbamid — Hydroxycarbamide Paediatric dispersible tablets will be provided in the form of film-coated dispersible tablets containing 50 mg of hydroxycarbamide.
  The IMP will be administered as half-strength twice daily, based on the body weight of the patient.
  Other Names: Hydroxyurea

SUMMARY:
The purpose of this interventional, phase II, national, multicentric, non-randomised, open-label study is to evaluate the pharmacokinetics (PK), efficacy and safety of Hydroxycarbamide Paediatric dispersible tablets with a twice daily dosing regimen in children with Sickle Celle Disease between 9 months to 11 years of age.

Participants will:

* Take Hydroxycarbamide twice a day every day for 12 months
* Visit the clinic at screening, baseline, 1, 3, 6, 9 and 12 months

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent, signed and dated by both parents or by the legally acceptable representative(s) of the children, and, if possible, assent from the children,
* HbSS or HbSβ0 SCD,
* Aged between 9 months and 11 years old,
* Hydroxycarbamide naïve,
* Parent(s) or legally acceptable representative(s) capable of communicating with the investigator and understanding the requirements and constraints of the study protocol and willing to comply with the study requirements,
* Contraception criterion, if applicable: for patients who are sexually active
* Affiliated to a social security plan or beneficiary of a similar insurance plan,
* Patient must meet the following laboratory values : Absolute Neutrophil Count ≥ 1.0x109/L, Platelets ≥ 75x109/L and Haemoglobin (Hgb) > 5.5 g/dL,
* Transcranial Doppler (TCD) in the last 12 months indicating low risk for stroke is required for children over 18 months of age.

Exclusion Criteria:

* Participation in any other clinical study for any other pharmaceutical product within 4 weeks preceding the inclusion visit,
* Patients who have had chronic blood transfusion or transfusion in the last 3 months preceding the inclusion visit,
* Patients treated with other SCD-modifying therapies,
* Patient with a stage 3, 4 or 5 chronic kidney disease,
* Patients known to be infected with human immunodeficiency virus, hepatitis B virus, or hepatitis C virus,
* Known hypersensitivity or allergy to the excipients,
* Any surgical or medical condition or any significant illness that, in the opinion of the investigator, constitutes a risk or a contraindication to the participation of the patient to the study, or that may interfere with the objectives, conduct or evaluation of the study,
* Female patients who are pregnant or lactating,
* Any documented history of a clinical stroke or intracranial haemorrhage, or an uninvestigated neurologic finding within the past 12 months.

Ages: 9 Months to 11 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 50 (Estimated)
Dates: Start 2025-01-21 (Actual); Primary Completion 2027-02 (Estimated); Study Completion 2027-02 (Estimated)

PRIMARY OUTCOMES:
Evaluate the PK exposure for Hydroxycarbamide Paediatric dispersible tablets administered BID through area under the curve (AUC) | 1, 3, 6, 9 and 12 months after treatment initiation
Evaluate the PK exposure for Hydroxycarbamide Paediatric dispersible tablets administered BID through time to obtain the maximum concentration (Tmax) | 1, 3, 6, 9 and 12 months after treatment initiation
Evaluate the PK exposure for Hydroxycarbamide Paediatric dispersible tablets administered BID through maximum plasma concentration (Cmax) | 1, 3, 6, 9 and 12 months after treatment initiation

SECONDARY OUTCOMES:
Absolute mean change from baseline in HbF levels | Baseline, 3, 6, 9 and 12 months after treatment initiation
HC plasma concentrations and HbF levels | Baseline, 3, 6, 9 and 12 months after treatment initiation
Daily AUC (AUC0-24h) at maintenance dose derived from the final PPK model | Baseline, 3, 6, 9 and 12 months after treatment initiation
Proportion of patients with a relative difference in Cmax ≥ 30% from BID maintenance dose relative to the one simulated on a once daily regimen giving an equivalent AUC0-24h. | Baseline, 3, 6, 9 and 12 months after treatment initiation
Absolute mean change from baseline in haematological parameters | Baseline,1, 3, 6, 9 and 12 months after treatment initiation
Acceptability score based on a hedonic face scale evaluated by the child from 3 years old | 3 months after treatment initiation
Acceptability score based on a 5-point Likert scale evaluated by the parent(s) or legally acceptable representative(s) | 3 months after treatment initiation
Distribution of the scores related to the ease of using the administration kit for treatment administration to the child based on a 5-point Likert scale evaluated by the parent(s) or legally acceptable representative(s) | 3 months after treatment initiation
  Score 1 : very difficult to score 5 : very easy
Compliance with Hydroxycarbamide Paediatric dispersible tablets administered BID by treatment unit accountability calculated by the pharmacy (patient will bring the kits with used and unused bottles to the pharmacy at each visit) | Baseline, 1, 3, 6, 9, 12 months after treatment initiation
Number of SCD events occurring during the study | Baseline, 1, 3, 6, 9, 12 months after treatment initiation
Number of adverse events (AEs) and percentage of patients reporting at least one AE | Baseline, 1, 3, 6, 9, 12 months after treatment initiation

CONTACTS AND LOCATIONS:
Overall Officials: Josephine Brice, MD, Principal Investigator — Hôpital Necker-Enfants Malades
Locations (6):
- France (5):
  - Centre Hospitalier Intercommunal Créteil, Créteil
  - GHEF- Site de Marne-la-Vallée, Jossigny
  - Hôpital Bicêtre, Le Kremlin-Bicêtre
  - Institut d'Hématologie et d'oncologie pédiatrique - IHOPe, Lyon
  - Hôpital Necker-Enfants malades, Paris
- Centre hospitalier de Cayenne, Cayenne, French Guiana

IPD SHARING:
Plan to Share IPD: No